CLINICAL TRIAL: NCT05356494
Title: Comparisons Effects of Postural Drainage and Positive Expiratory Pressure Technique in Community Acquired Pneumonia.
Brief Title: Postural Drainage and PEP Technique in Community Acquired Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0318 M Ahmad
Record Dates: First submitted 2022-04-28; First posted 2022-05-02 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Community-acquired Pneumonia
Keywords: Pneumonia,; Postural Drainage; Positive Expiratory Pressure
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia | interventions — Drainage, Postural; Positive-Pressure Respiration

STUDY DESIGN:
Intervention Model Description: The study concluded that both techniques are effective in improving oxygen saturation and reported statistically significant differences, but no other parameter was statistically improved.
Who Masked: Participant
Masking Description: The results of the study are in accordance with current study but for improvement in oxygen saturation. However, other variables of ABGs did not show significant improvement after both techniques in community acquired pneumonia patients. In contrast to previous study, the techniques are only effective for improving saturation in patients with community acquired pneumonia.
  single blinded study only participant blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postural drainage (Experimental): (Group A will be treated with postural drainage)
  Interventions: Other: Postural drainage
- positive expiratory pressure technique (Experimental): (Group B will be treated with positive expiratory pressure technique).
  Interventions: Other: Positive expiratory pressure

INTERVENTIONS:
Other: Postural drainage — (Group A will be treated with postural drainage)
  Arms: postural drainage
Other: Positive expiratory pressure — (Group B will be treated with positive expiratory pressure technique).
  Arms: positive expiratory pressure technique

SUMMARY:
Community-acquired pneumonia is acquired outside the hospital. Postural drainage is the positioning of a patient with an involved lung segment such that gravity has a maximal effect of facilitating the drainage of Broncho-pulmonary secretions from the tracheobronchial tree. It is based on the concept of gravity-assisted mobilization of secretions and transports it for removal. The objective of the study to find the effect of postural drainage and positive expiratory pressure techniques (PEP) to improve the air way clearance and breathing in pneumonia patients. This study will be a RCT and will be conducted in Services Hospital. The study will be completed within the duration of six month. Consecutive sampling study technique will be used to collect the data. The sample size of 46 patients will be taken. Patients will be divided into two groups. (Group A will be treated with postural drainage and Group B will be treated with positive expiratory pressure technique). Outcome measure will be taken on Pulse oximeter, incentive spirometer and chest X- Ray. A regular follow up visits to department and a final assessment was made at the end of four week. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro- Wilk test, it will be decided either parametric or non-parametric test will be use within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with community acquired pneumonia.
* Clinically stable patients.
* Both genders
* Age 30 to 70 years

Exclusion Criteria:

* Presence of any genetic disorders (cystic fibrosis).
* Recent spinal / chest surgery
* Cardiac issues
* Fractures of vertebra caused by osteoporosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
INCENTIVE SPIROMETER | 1 Last week
  An incentive spirometer is a handheld device that helps your lungs recover after a surgery or lung illness. When you breathe from an incentive spirometer, a piston rises inside the device and measures the volume of your breath. A healthcare provider can set a target breath volume for you to hit.
OXYGEN SATURATION | 1 Last week
  Oxygen saturation, or "O2 sates," indicates that amount of oxygen traveling through your body with your red blood cells. Normal oxygen saturation is usually between 95% and 100% for most health.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, MS.CPPT, Principal Investigator — Riphah International University
Locations (1):
- Services Hospital, Lahore., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li L, Qin L, Xu Z, Yin Y, Wang X, Kong B, Bai J, Lu Y, Fang Z, Song Q, Cao K, Liu D, Wang G, Xu Q, Fang X, Zhang S, Xia J, Xia J. Using Artificial Intelligence to Detect COVID-19 and Community-acquired Pneumonia Based on Pulmonary CT: Evaluation of the Diagnostic Accuracy. Radiology. 2020 Aug;296(2):E65-E71. doi: 10.1148/radiol.2020200905. Epub 2020 Mar 19. PMID 32191588
- [Background] Ouyang X, Huo J, Xia L, Shan F, Liu J, Mo Z, Yan F, Ding Z, Yang Q, Song B, Shi F, Yuan H, Wei Y, Cao X, Gao Y, Wu D, Wang Q, Shen D. Dual-Sampling Attention Network for Diagnosis of COVID-19 From Community Acquired Pneumonia. IEEE Trans Med Imaging. 2020 Aug;39(8):2595-2605. doi: 10.1109/TMI.2020.2995508. PMID 32730212
- [Background] Metlay JP, Waterer GW. Treatment of Community-Acquired Pneumonia During the Coronavirus Disease 2019 (COVID-19) Pandemic. Ann Intern Med. 2020 Aug 18;173(4):304-305. doi: 10.7326/M20-2189. Epub 2020 May 7. PMID 32379883
- [Background] Wang Z, Xiao Y, Li Y, Zhang J, Lu F, Hou M, Liu X. Automatically discriminating and localizing COVID-19 from community-acquired pneumonia on chest X-rays. Pattern Recognit. 2021 Feb;110:107613. doi: 10.1016/j.patcog.2020.107613. Epub 2020 Aug 26. PMID 32868956
- [Background] Pernica JM, Harman S, Kam AJ, Carciumaru R, Vanniyasingam T, Crawford T, Dalgleish D, Khan S, Slinger RS, Fulford M, Main C, Smieja M, Thabane L, Loeb M. Short-Course Antimicrobial Therapy for Pediatric Community-Acquired Pneumonia: The SAFER Randomized Clinical Trial. JAMA Pediatr. 2021 May 1;175(5):475-482. doi: 10.1001/jamapediatrics.2020.6735. PMID 33683325
- [Background] Waseem MH, Lasi FF, Valecha J, Samejo B, Sangrasi SA, Ali SM. Effectiveness of Chest Physiotherapy in Cerebrovascular Accident Patients With Aspiration Pneumonia. Journal of Modern Rehabilitation. 2021;15(1):47-52.
- [Background] Ryrso CK, Faurholt-Jepsen D, Ritz C, Pedersen BK, Hegelund MH, Dungu AM, Sejdic A, Lindegaard B, Krogh-Madsen R. The impact of physical training on length of hospital stay and physical function in patients hospitalized with community-acquired pneumonia: protocol for a randomized controlled trial. Trials. 2021 Aug 28;22(1):571. doi: 10.1186/s13063-021-05503-2. PMID 34454594
- [Background] Nair GB, Niederman MS. Updates on community acquired pneumonia management in the ICU. Pharmacol Ther. 2021 Jan;217:107663. doi: 10.1016/j.pharmthera.2020.107663. Epub 2020 Aug 15. PMID 32805298
- [Background] Leemans G, Belmans D, Van Holsbeke C, Becker B, Vissers D, Ides K, Verhulst S, Van Hoorenbeeck K. The effectiveness of a mobile high-frequency chest wall oscillation (HFCWO) device for airway clearance. Pediatr Pulmonol. 2020 Aug;55(8):1984-1992. doi: 10.1002/ppul.24784. Epub 2020 Apr 22. PMID 32320537